CLINICAL TRIAL: NCT03384368
Title: A Modified Placement of Two Additional Pedicle Screws at the Fracture Level for the Treatment of Thoracolumbar Burst Fractures--a Study Protocol of a Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2017-08-115
Record Dates: First submitted 2017-12-05; First posted 2017-12-27 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Posterior Short-segment Pedicle Instrumentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screw-Distraction (SD) group (Placebo Comparator): six pedicle screws were implanted firstly, then distraction was achieved.
  Interventions: Device: fractured level screws-distraction
- Distraction-Screw (DS) group (Experimental): four pedicle screws were implanted firstly, then distraction was achieved, two additional screws were introduced at the fracture level at last.
  Interventions: Device: fractured level screws-distraction

INTERVENTIONS:
Device: fractured level screws-distraction — four pedicle screws were implanted into the upper vertebra and the lower vertebral body of the fractured vertebra. Then, immediate reduction and decompression were achieved by applying distraction of rod. Finally, two additional screws were introduced at fracture level

SUMMARY:
Controversies exist about the best treatment of burst fractures of the thoracolumbar spine. Adding screws in fractured segment has been proved in many literatures that can improve construct stiffness but sometimes aggravate the trauma of fractured vertebra. Therefore, we are eager to find an optimized placement of two additional pedicle screws at the fracture level for the treatment of thoracolumbar burst fractures. This is the first randomised controlled study investigating efficacy of diverse orders of pedicle screws placement and will provide recommendations for treating patients with thoracolumbar burst fractures.

DETAILED DESCRIPTION:
A blinded randomised controlled trial (blinding for the patient and statistician, rather than for the clinician and researcher) will be conducted. A total of seventy patients with single thoracolumbar AO type A3 or A4 fractures who are candidates for application of short-segment pedicle screws of fractured vertebrae will be randomly allocated to either the DS group (distraction-screws ) or the SD group (screws-distraction) at a ratio of 1: 1. The primary clinical outcome measures are compression ratio of anterior border of vertebral body height, depth of nail into injured vertebrae and kyphosis (Cobb) angle. Secondary clinical outcome measures are complications, Visual Analogue Scale (VAS) of back and leg pain, neurological function, operating time, intraoperative blood loss, Japanese Orthopaedic Association (JOA) scores and Oswestry Disability Index. These parameters will be evaluated preoperatively, intraoperatively, on day 3 postoperatively and then at 1, 3, 6, 12 and 24 months postoperatively.

ELIGIBILITY:
Inclusion criteria

1. 18 years of age or above.
2. single thoracolumbar burst fractures
3. AO type A3 or A4 fractures
4. Thoracolumbar Injury Classification and Severity Score (TLICS) of more than 4 and duration of < 2 weeks
5. application of posterior short-segment pedicle screws instrumentation at the fracture level Exclusion criteria

1. previous pedicle instrumentation at the same level 2. multi-segmental thoracolumbar fractures or not AO type A3 or A4 are found 3. pregnancy 4. active infection or surgical site of the previous infection 5. planned emigration abroad within 2 years after inclusion 6. suffering from illness or long-term use of certain drugs affecting the stability of the spinal environment, such as metabolic bone disease, spinal tuberculosis and so on 7. the current use of anticoagulant (such as warfarin) or postoperative heparin for more than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
compression ratio change of anterior border of vertebral body height | preoperatively, intraoperatively, on day 3 postoperatively and then at 1, 3, 6, 12 and 24 months postoperatively
  using X-ray fluorescence
Depth of nail into injured vertebrae | at postoperation immediately
  using X-ray fluorescence
Kyphosis (Cobb) angle change | preoperatively, intraoperatively, on day 3 postoperatively and then at 1, 3, 6, 12 and 24 months postoperatively
  using X-ray fluorescence

SECONDARY OUTCOMES:
Operative time | right after surgery
  Unit of Measure is hour
intraoperative blood loss | right after surgery
  Unit of Measure is ml
Complications | at postoperation immediately, 1, 3 and 6 months, and at 1 and 2 years postoperatively.
  Pedicle fractures, intraoperative pars fractures, postoperative infection, deep venous thrombosis, nerve injury, and any other direct or indirect surgical complications will be recorded.
pain degree of back and lower limb | preoperatively, on day 3 postoperatively and then at 1, 3, 6, 12 and 24 months postoperatively.
  The pain degree of back and lower limb during follow-up will be assessed by the VAS of back pain and VAS of leg pain
Oswestry Disability Index (ODI) change | preoperatively, on day 3 postoperatively and then at 1, 3, 6, 12 and 24 months postoperatively
  The Oswestry Disability Index (ODI) will be asssessed by questionnaire
The Japanese Orthopaedic Association (JOA) scores | preoperatively and postoperatively including day 3 and then 1, 3, 6, 12 and 24 months
  Functional improvement is expressed by the rate of recovery of the JOA scores
The American Spinal Injury Association (ASIA) impairment scale | preoperatively, on day 3 postoperatively and then at 1, 3, 6, 12 and 24 months postoperatively
  Spinal Injury was assessed using ASIA

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Hu ZC, Li XB, Feng ZH, Wang JQ, Gong LF, Xuan JW, Fu X, Jiang BJ, Wu L, Ni WF. Modified pedicle screw placement at the fracture level for treatment of thoracolumbar burst fractures: a study protocol of a randomised controlled trial. BMJ Open. 2019 Jan 28;9(1):e024110. doi: 10.1136/bmjopen-2018-024110. PMID 30696677